CLINICAL TRIAL: NCT03828526
Title: Effectiveness of High Fidelity Simulation for Safety in the Medication Process in Intensive Care: Randomized Clinical Trial
Brief Title: Effectiveness of High Fidelity Simulation for Safety in the Medication Process in Intensive Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Marcia Cristina da Silva Magro, Principal Investigator, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: U1111-1227-7554
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Learning Process in Nursing Graduation; Compliant Behavior
Keywords: Patient Safety; Medication Errors; Critical Care; Nursing Education; High Fidelity Simulation Training
MeSH Terms: conditions — Cooperative Behavior

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Fidelity Simulation (Experimental): Students will be exposed to the intensive care setting where they will have to solve issues related to general nursing care, including the stages of the medication process that involve the nurses' performance and their complexity.
  During the experience of the scenario will be provoked external factors, such as telephone ringing, visit of the professional of the infection commission, to evaluate the reactions of the student and the strategies adopted to minimize the occurrence of adverse events against such external factors.
  Subsequently, they will participate in the debriefing, where they will be reflected on the positives and those that should be adjusted to promote safer nursing care related to drug administration.
  Interventions: Other: High Fidelity Simulation
- Traditional teaching strategy (Active Comparator): Participants will be submitted to an expository-dialogue class, which will be given based on the recent literature and subdivided into the following axes: 1) patient safety; 2) medication process; 3) adverse drug events; 4) the critical patient in intensive care and its specificities. Afterwards, students will be directed to an environment with an anatomical piece for drug preparation and administration training.
  Interventions: Other: Traditional teaching strategy

INTERVENTIONS:
Other: High Fidelity Simulation — Teaching strategy based on high fidelity simulation, which simulates the reality of health care to promote meaningful learning.
  Arms: High Fidelity Simulation
Other: Traditional teaching strategy — Classroom-based strategy
  Arms: Traditional teaching strategy

SUMMARY:
Nursing plays an important role in the medication process in intensive care units. The application of active methodologies guided by the simulation strategy can help in the formation of qualified professionals and in the safer promotion of health care. The objectives to evaluate the effectiveness of the high fidelity simulation applied to nursing students in the process of administering drugs to critical patients in the intensive care setting; evaluate knowledge acquisition, satisfaction and self-confidence after the simulation. This is a prospective, single-blinded, controled clinical trial, with a quantitative approach. The sample will be composed of nursing students who are attending or have completed the discipline of critical care. The students will be randomized electronically to the experimental group, whose intervention will be guided by the high fidelity simulation method and, to the control group, the handling of static dummies / traditional teaching will be adopted as teaching strategy. Both strategies will emphasize the safety process during medication administration to critical patients hospitalized in the intensive care unit and will have an expository class dialogued prior to the intervention. Pre and post-tests will be applied at different times to evaluate the evolution of the level of knowledge and its retention and also, scales of satisfaction and self-confidence in learning. Descriptive and inferential statistics will be performed, as appropriate. It is believed that students submitted to simulation will have the opportunity to better consolidate knowledge during the training process, improve clinical and critical thinking, and decision-making, which will positively influence the safety of critically ill patients of the intensive care unit.

DETAILED DESCRIPTION:
Objective

To evaluate the effectiveness of the high fidelity simulation for learning related to the drug preparation and administration process in the scenario of critical patient care in the cognitive, psychomotor and affective domains for undergraduate students of the nursing course.

Hypothesis of the study

Null hypothesis

There will be no difference between learning through high fidelity simulation and traditional teaching / low fidelity simulation.

Alternative hypothesis

The high fidelity simulation strategy improves the performance of nursing students in drug administration more significantly when compared to traditional teaching / low fidelity simulation.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled in the undergraduate nursing course of a public university in Brazil; Students coursing or who have completed critical care discipline.

Exclusion Criteria:

* Students with previous training in health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Previous knowledge about the preparation and administration of intravenous drugs in intensive care (pre-test) | Questionnaire application prior to the intervention (pre-test)
  It will be measured by applying a "Knowledge Questionnaire" consisting of 5 objective questions to study participants. The minimum score on the test will be 0 points (worst score) and the maximum score will be 100 points (best score).
Knowledge about the preparation and administration of intravenous drugs in intensive care (post-test) | Questionnaire application immediately after the intervention (post-test)
  It will be measured by applying a "Knowledge Questionnaire" consisting of 5 objective questions to study participants. The minimum score on the test will be 0 points (worst score) and the maximum score will be 100 points (best score).
Knowledge about the preparation and administration of intravenous drugs in intensive care (1st retention) | Questionnaire application one month after intervention (1st retention)
  It will be measured by applying a "Knowledge Questionnaire" consisting of 5 objective questions to study participants. The minimum score on the test will be 0 points (worst score) and the maximum score will be 100 points (best score).
Knowledge about the preparation and administration of intravenous drugs in intensive care (2nd retention) | Questionnaire application three months after intervention (1st retention)
  It will be measured by applying a "Knowledge Questionnaire" consisting of 5 objective questions to study participants. The minimum score on the test will be 0 points (worst score) and the maximum score will be 100 points (best score).

SECONDARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning | The scale will be applied in two distinct times: Time 1 - before the intervention; Time 2 - immediately after the intervention.
  It will be measured through the application of the "Student Satisfaction and Self-Confidence in Learning" scale, composed of 13 items. Each item should be marked on a scale from 1 (worst score) to 5 (best score), where 1 - strongly disagree with the statement; 2 - I disagree with the statement; 3 - I do not agree or disagree; 4 - I agree with the statement; 5 - strongly agree with the statement.
Perceived gains from high fidelity simulation | The scale will be applied immediately after the intervention.
  It will be measured through the application of the "High-fidelity simulation gains on nursing education" scale, composed of 26 items related to the skills developed through the simulation strategy. Each item should be marked on a scale from 1 (worst score) to 5 (best score), where 1 - I get worse; 2 - remained the same; 3 - I have improved little; 4 - I have improved considerably; 5 - I have improved immensely.

CONTACTS AND LOCATIONS:
Overall Officials: Marcia CS Magro, PhD, Study Director — University of Brasilia
Locations (1):
- Breno de Sousa Santana, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams AJ, Wasson EA, Admire JR, Pablo Gomez P, Babayeuski RA, Sako EY, Willis RE. A Comparison of Teaching Modalities and Fidelity of Simulation Levels in Teaching Resuscitation Scenarios. J Surg Educ. 2015 Sep-Oct;72(5):778-85. doi: 10.1016/j.jsurg.2015.04.011. Epub 2015 May 20. PMID 26002536
- [Background] Bingham AL, Sen S, Finn LA, Cawley MJ. Retention of advanced cardiac life support knowledge and skills following high-fidelity mannequin simulation training. Am J Pharm Educ. 2015 Feb 17;79(1):12. doi: 10.5688/ajpe79112. PMID 25741028
- [Background] Choi I, Lee SM, Flynn L, Kim CM, Lee S, Kim NK, Suh DC. Incidence and treatment costs attributable to medication errors in hospitalized patients. Res Social Adm Pharm. 2016 May-Jun;12(3):428-37. doi: 10.1016/j.sapharm.2015.08.006. Epub 2015 Aug 20. PMID 26361821
- [Background] Cortegiani A, Russotto V, Montalto F, Iozzo P, Palmeri C, Raineri SM, Giarratano A. Effect of High-Fidelity Simulation on Medical Students' Knowledge about Advanced Life Support: A Randomized Study. PLoS One. 2015 May 8;10(5):e0125685. doi: 10.1371/journal.pone.0125685. eCollection 2015. PMID 25955760
- [Background] Institute of Medicine (US) Committee on Quality of Health Care in America; Kohn LT, Corrigan JM, Donaldson MS, editors. To Err is Human: Building a Safer Health System. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK225182/ PMID 25077248
- [Background] Marvanova M, Henkel PJ. Collaborating on medication errors in nursing. Clin Teach. 2018 Apr;15(2):163-168. doi: 10.1111/tct.12655. Epub 2017 Apr 24. PMID 28436158
- [Background] Negri EC, Mazzo A, Martins JCA, Pereira GA Junior, Almeida RGDS, Pedersoli CE. Clinical simulation with dramatization: gains perceived by students and health professionals. Rev Lat Am Enfermagem. 2017 Aug 3;25:e2916. doi: 10.1590/1518-8345.1807.2916. PMID 28793125
- [Background] Renata Grou Volpe C, Moura Pinho DL, Morato Stival M, Gomes de Oliveira Karnikowski M. Medication errors in a public hospital in Brazil. Br J Nurs. 2014 Jun 12-25;23(11):552, 553-9. doi: 10.12968/bjon.2014.23.11.552. PMID 24933543